CLINICAL TRIAL: NCT04781738
Title: Functional Capacity and Quality of Life in Patients With Vascular Ring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, l_bentur, Principal Investigator, Rambam Health Care Campus
Other Study IDs: RMB-0218-17
Record Dates: First submitted 2021-02-21; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Vascular Ring
Keywords: Cardiopulmonary exercise testing,; Double aortic arch
MeSH Terms: conditions — Vascular Ring | interventions — Exercise Test; Walk Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with history of vascular ring who didn't have corrective surgery: patients with history of vascular ring who didn't have corrective surgery
  Interventions: Diagnostic Test: Cardiopulmonary exercise test
- patients with history of vascular ring who underwent corrective surgery: patients with history of vascular ring who underwent corrective surgery
  Interventions: Diagnostic Test: Cardiopulmonary exercise test

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test — CPET using a cycle ergometer (COSMED, Rome, Italy) beginning with no resistance warmup lasting 1-3 minutes followed with an incrementing resistance adapted to the patient's functional capacities according to the examiner's free judgment by successive stages
  Six minute walk test - patients will be instructed to walk as far as possible for six minutes in a 30-meter long enclosed corridor with a flat and hard surface, marked at every meter. Meters will be calculated at the end of the test.
  SF-36 is a questionnaire that contains eight domains - physical functioning (10 items); role limitations due to physical functioning (4 items); role limitations due to emotional problems (3 items); energy and vitality (4 items); mental health (5 items); social functioning (2 items); bodily pain (2 items); and general health perceptions (5 items).
  Scores are summed for each domain and were transformed into scores of between 0 (worst possible health state) to 100 (best possible health state).
  Other Names: 6 minute walk test; quality of life questionnaire (sf-36)

SUMMARY:
To investigate the long term functional capacity and quality of life of patients with a history of vascular ring whether they did or did not have corrective surgery. Patients will perform pulmonary function test, 6 minute walk test, cardiopulmonary exercise test and will fill a quality of life questionnaire.

DETAILED DESCRIPTION:
Vascular rings are congenital vascular anomalies of the aortic arch that compress the esophagus and the trachea. The most common vascular rings are double aortic arch and right aortic arch with left ligamentum. Pulmonary artery sling is less common. Another cause of tracheal compression occurring only in infants is the innominate artery compression syndrome. When patients are symptomatic, surgical correction should be performed.

data regarding long term functional capacity and quality of life is lacking. our aim is to investigate the long term functional capacity and quality of life of patients with history of vascular ring whether they did or did not have corrective surgery.

Methods: a prospective study evaluating functional capacity and quality of life the patients will perform pulmonary function test, 6 minute walk test, cardiopulmonary exercise test and will fill a quality of life questionnaire (sf-36).

ELIGIBILITY:
Inclusion Criteria:

* patients with history of vascular ring

Exclusion Criteria:

* refusal to participate
* inability to complete cardiopulmonary testing

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with history of vascualr ring
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Measured continuously during 15 minutes of the exercise test (CPET)
  Oxygen uptake evaluated by cardiopulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
Six minute walk test | Six minutes of evaluation, completed pre cardiopulmonary exercise test (CPET)
  The distance gained after six minute of habitual walking.
Quality of life - SF-36 | Five minutes of evaluation, completed pre cardiopulmonary exercise test (CPET)
  The calculated result of SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Principal Investigator — Head of Pediatric Pulmonary Institute
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nir V, Bentur L, Zucker-Toledano M, Gur M, Adler Z, Hanna M, Toukan Y, Masarweh K, Hakim F, Bar-Yoseph R. Functional capacity and quality of life in patients with vascular ring. Pediatr Pulmonol. 2022 Dec;57(12):2946-2953. doi: 10.1002/ppul.26112. Epub 2022 Sep 14. PMID 35971243